CLINICAL TRIAL: NCT04157868
Title: The Impact of Early rhBNP on Myocardial Work in Patients With Anterior ST-segment Elevation Myocardial Infarction After Percutaneous Coronary Intervention
Brief Title: Early rhBNP on Myocardial Work in Patients With STEMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EARLY MYO-myocardial work
Record Dates: First submitted 2019-11-05; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: ST-Segment Elevated Myocardial Infarction
Keywords: ST-Segment Elevated Myocardial Infarction; rhBNP; non-invasive myocardial work

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhBNP (Experimental): rhBNP intra-coronary injection 1.5 ug/kg loading dose, with intravenous injection 0.0075-0.01 ug/kg/min persistent for 72 hour.
  Interventions: Drug: rhBNP
- Control (Placebo Comparator): Saline intra-coronary injection 0.15ml/kg loading dose, with same intravenous injection speed for 72 hour after randomization.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: rhBNP — rhBNP intra-coronary injection 1.5 ug/kg loading dose, with intravenous injection 0.0075-0.01 ug/kg/min persistent for 72 hour.
  Arms: rhBNP
Drug: Control — Saline intra-coronary injection 0.15ml/kg loading dose, with same intravenous injection speed for 72 hour.
  Arms: Control

SUMMARY:
The study intends to evaluate the efficacy of early rhBNP on myocardial work in patients with anterior ST-segment elevation myocardial infarction after percutaneous coronary intervention

ELIGIBILITY:
Inclusion Criteria:

* 1. Anterior myocardial infarct (anterior myocardial infarct is defined as persistent chest pain for 30 mins at least, with ST-segment elevation of at least 0.2 mV in two or more contiguous precordial leads) within 12 hours after onsets of symptom;

  2. No contraindication for rhBNP;

  3. Left anterior descending (LAD) as culprit vessel, with TIMI 0-1 grade.

Exclusion Criteria:

* 1.Cardiogenic shock (systolic BP <90mmHg after fluid infusion or systolic BP<100mmHg after vasoactive drugs);

  2. History of myocardial infarct;

  3.Severe arrhythmia: with III degree A-V block ,atrial fibrillation,ventricular fibrillation,ventricular tachycardia;

  4. Any history of severe renal or hepatic dysfunction (hepatic failure, cirrhosis, portal hypertension or active hepatitis); neutropenia or thrombocytopenia; known acute pancreatitis;

  5. Pregnant or lactating;

  6. life expectancy≤12 months;

  7. Inability to follow the protocol and comply with follow-up requirements or any other reason the investigator feels would place the patient at increased risk;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-11-30 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Global myocardial work efficiency by echocardiography | 30 days after PCI
  Echocardial myocardial work (MW) may identify early abnormalities in left ventricular(LV) function and may establish a more sensitive index for early stage LV dysfunction.Global MW was quantified by calculating the rate of regional shortening by differentiation of the strain tracing and multiplying by instantaneous LV pressure. This instantaneous measure of power was this integrated over time to measure MW as a function of time during systole (time interval from mitral valve closure through to mitral valve opening). During LV ejection, segments were analyzed for wasted work (WW) and/or constructive work (CW), with global values determined as the averages of all segmental values and displayed on the LV pressure-strain loop diagram.
  Global myocardial work efficiency (GWE; %), constructive MW divided by the sum of CW and WW, expressed as a percentage.

SECONDARY OUTCOMES:
Global myocardial work index by echocardiography | Day 1, 7, 30 after PCI
  Global myocardial work index (GWI): total work within the area of the LV PSL calculated frommitral valve closure to mitral valve opening.
Global myocardial constructive work by echocardiography | Day 1, 7, 30 after PCI
  Global myocardial constructive work (mm Hg %), an estimate of the work performed by the LV segments consisting of shortening during systole plus lengthening in isovolumic relaxation.
Global myocardial waste work by echocardiography | Day 1, 7, 30 after PCI
  Global myocardial waste work (mm Hg %), an estimate of negative work of the LV segments consisting of myocardial lengthening during systole plus any shortening during isovolumic relaxation.
Clinical Outcomes | 30 days after PCI
  Compound endpoints of all cause death, non-fatal reinfarction, heart failure, and stroke;

CONTACTS AND LOCATIONS:
Overall Officials: Song Ding, MD,Ph.D., Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schwartz BG, Kloner RA. Coronary no reflow. J Mol Cell Cardiol. 2012 Apr;52(4):873-82. doi: 10.1016/j.yjmcc.2011.06.009. Epub 2011 Jun 21. PMID 21712046
- [Background] Niccoli G, Burzotta F, Galiuto L, Crea F. Myocardial no-reflow in humans. J Am Coll Cardiol. 2009 Jul 21;54(4):281-92. doi: 10.1016/j.jacc.2009.03.054. PMID 19608025
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Background] Kehat I, Molkentin JD. Molecular pathways underlying cardiac remodeling during pathophysiological stimulation. Circulation. 2010 Dec 21;122(25):2727-35. doi: 10.1161/CIRCULATIONAHA.110.942268. No abstract available. PMID 21173361
- [Background] Postma S, Dambrink JH, Gosselink AT, Ottervanger JP, Kolkman E, Ten Berg JM, Suryapranata H, van 't Hof AW. The influence of system delay on 30-day and on long-term mortality in patients with anterior versus non-anterior ST-segment elevation myocardial infarction: a cohort study. Open Heart. 2015 Apr 10;2(1):e000201. doi: 10.1136/openhrt-2014-000201. eCollection 2015. PMID 25893101
- [Background] Wu GF, Wykrzykowska JJ, Rana JS, Pinto DS, Gibson CM, Li J, Sellke FW, Laham RJ. Effects of B-type natriuretic peptide (nesiritide) on coronary epicardial arteries, systemic vasculature and microvessels. J Invasive Cardiol. 2008 Feb;20(2):76-80. PMID 18252972
- [Background] Sjoli B, Orn S, Grenne B, Ihlen H, Edvardsen T, Brunvand H. Diagnostic capability and reproducibility of strain by Doppler and by speckle tracking in patients with acute myocardial infarction. JACC Cardiovasc Imaging. 2009 Jan;2(1):24-33. doi: 10.1016/j.jcmg.2008.10.007. PMID 19356529
- [Background] Shimoni S, Gendelman G, Ayzenberg O, Smirin N, Lysyansky P, Edri O, Deutsch L, Caspi A, Friedman Z. Differential effects of coronary artery stenosis on myocardial function: the value of myocardial strain analysis for the detection of coronary artery disease. J Am Soc Echocardiogr. 2011 Jul;24(7):748-57. doi: 10.1016/j.echo.2011.03.007. Epub 2011 Apr 20. PMID 21511433
- [Background] Hubert A, Le Rolle V, Leclercq C, Galli E, Samset E, Casset C, Mabo P, Hernandez A, Donal E. Estimation of myocardial work from pressure-strain loops analysis: an experimental evaluation. Eur Heart J Cardiovasc Imaging. 2018 Dec 1;19(12):1372-1379. doi: 10.1093/ehjci/jey024. PMID 29529181
- [Background] Donal E, Bergerot C, Thibault H, Ernande L, Loufoua J, Augeul L, Ovize M, Derumeaux G. Influence of afterload on left ventricular radial and longitudinal systolic functions: a two-dimensional strain imaging study. Eur J Echocardiogr. 2009 Dec;10(8):914-21. doi: 10.1093/ejechocard/jep095. Epub 2009 Aug 7. PMID 19666722
- [Background] Edwards NFA, Scalia GM, Shiino K, Sabapathy S, Anderson B, Chamberlain R, Khandheria BK, Chan J. Global Myocardial Work Is Superior to Global Longitudinal Strain to Predict Significant Coronary Artery Disease in Patients With Normal Left Ventricular Function and Wall Motion. J Am Soc Echocardiogr. 2019 Aug;32(8):947-957. doi: 10.1016/j.echo.2019.02.014. Epub 2019 Apr 28. PMID 31043359
- [Background] Masci PG, Marinelli M, Piacenti M, Lorenzoni V, Positano V, Lombardi M, L'Abbate A, Neglia D. Myocardial structural, perfusion, and metabolic correlates of left bundle branch block mechanical derangement in patients with dilated cardiomyopathy: a tagged cardiac magnetic resonance and positron emission tomography study. Circ Cardiovasc Imaging. 2010 Jul;3(4):482-90. doi: 10.1161/CIRCIMAGING.109.934638. Epub 2010 May 12. PMID 20463209
- [Background] Duchenne J, Turco A, Unlu S, Pagourelias ED, Vunckx K, Degtiarova G, Bezy S, Cvijic M, Nuyts J, Claus P, Rega F, Gheysens O, Voigt JU. Left Ventricular Remodeling Results in Homogenization of Myocardial Work Distribution. Circ Arrhythm Electrophysiol. 2019 May;12(5):e007224. doi: 10.1161/CIRCEP.118.007224. PMID 31023060
- [Background] Boe E, Russell K, Eek C, Eriksen M, Remme EW, Smiseth OA, Skulstad H. Non-invasive myocardial work index identifies acute coronary occlusion in patients with non-ST-segment elevation-acute coronary syndrome. Eur Heart J Cardiovasc Imaging. 2015 Nov;16(11):1247-55. doi: 10.1093/ehjci/jev078. Epub 2015 Apr 6. PMID 25851329